CLINICAL TRIAL: NCT06889662
Title: GEAM: Yield of GEnetic Testing in Arrhythmic Myocarditis
Brief Title: GEAM Study Aims At Assessing the Role of Genetic Testing in Patients with Arrhythmic Myocarditis.
Acronym: GEAM
Status: Recruiting | Type: Observational
Sponsor: Scientific Institute San Raffaele (Other)
Responsible Party: Principal Investigator, Giovanni Peretto, Medical Doctor, PhD, Principal Investigator, Scientific Institute San Raffaele
Other Study IDs: GEAM
Record Dates: First submitted 2025-02-06; First posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-02

CONDITIONS: Myocarditis; Ventricular Arrythmia
Keywords: Arrhythmogenic cardiomyopathy; Ventricular arrhythmias; Myocardial inflammation
MeSH Terms: conditions — Myocarditis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- VA+: with ventricular arrhythmias
- VA-: without ventricular arrhythmias

SUMMARY:
This study aims to answer multiple unsolved questions in the field of arrhythmic myocarditis.

* Improving the diagnostic work-up. While endomyocardial biopsy (EMB) and cardiac magnetic resonance (CMR) constitute the gold standard diagnostic techniques for myocarditis, the role of genetic testing is still unclear. Identifying the subset of patients with CGVs, will contribute to justifying the application of genetic testing in myocarditis.
* Generating models for risk prediction. Outcomes and arrhythmic risk stratification remain uncertain for myocarditis. Based on an advanced multimodal work-up, multiparametric risk scores may be created and subsequently validated, in order to predict the arrhythmic risk of specific myocarditis, especially in the case of CGVs.
* Identifying disease-specific and genotype-specific signatures. Genotype-phenotype associations are expected to benefit from a multimodal and multiparametric approach, in order to allow etiology-specific features in arrhythmic myocarditis. Most of the current signatures are limited to combined EMB-CMR studies. Signatures would likely benefit from implementing additional parameters, including arrhythmia features and myocardial inflammatory status.
* Tailoring treatment strategies. Transcriptional analysis will identify overexpressed genes associated with myocarditis and arrhythmias, representing a possible therapeutic target. A multimodal and multidisciplinary model will integrate phenotype, genotype, and transcriptional profile for a personalized treatment.

DETAILED DESCRIPTION:
Arrhythmic myocarditis is responsible for a significant proportion of out-of-hospital cardiac arrest and death in the young population. Although considered an uncommon feature, arrhythmias may present in myocarditis in both acute and chronic phase, leading to sudden cardiac death (SCD), especially in young males. Overall, the prevalence of undiagnosed myocarditis in post-mortem series ranges from 9% to 44%, involving 2% of infants, 5% of children, and 4-8% of athletes <40-year-old. Ventricular arrhythmias (VAs) are reported secondary to lymphocytic myocarditis. However, they are more commonly associated with giant cell myocarditis (GCM) and cardiac sarcoidosis (CS), with prevalence of 29% and 55%, respectively In addition, genetically-determined susceptibility might underlie arrhythmic myocarditis.

First, recent reports suggest that pathogenic variants in genes associated with nonischemic cardiomyopathies (NICM), hereby defined as cardiomyopathic gene variants (CGVs) are frequently found in patients with myocarditis proven by CMR and/or EMB, complicated by ventricular arrhythmias (VA). NICM constitute a heterogeneous group of diseases characterized by distinct structural and functional myocardial abnormalities in the absence of obstructive epicardial coronary artery disease. The main NICM overlapping with myocarditis are dilated (DCM) and arrhythmogenic cardiomyopathy (ACM).

Second, myocardial inflammation (M-Infl) has also been recently described in NICM complicated by arrhythmias. Preclinical data support a relevant role of M-Infl in the pathophysiology of AINICM, and its association with adverse outcomes.

Furthermore, there is a growing interest in transcriptomics in the setting of inflammatory and genetic cardiomyopathies. Cardiac transcriptome revealed specific subgroups of patients with early and overt DCM. In animal models of experimental autoimmune myocarditis, transcriptomics, transcriptomics allowed to depict the single-cell landscape of the cardiac immune cells in different phases of the disease. The addition of the cardiac transcriptome to the genotype and phenotype of patients increases the possibility for individualized medicine.

ELIGIBILITY:
Inclusion Criteria:

Patients with ventricular arrhythmias (VA+) and without (VA-)

* Diagnosis of myocarditis proven by EMB (ESC criteria) and/or CMR (updated Lake Louise criteria)
* Age ≥ 10 years
* Baseline ECG telemonitoring
* Written informed consent Healthy controls
* Provided a negative known history of myocarditis
* The sample must have been biobanked as part of the study IMMUNORADAR

Exclusion Criteria:

Patients with ventricular arrhythmias (VA+) and without (VA-)

* Obstructive coronary artery disease, or lack of coronary angiography/computed tomography (CT) scan in patients >40 years.
* Absent informed consent.

Ages: 10 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Statistical analyses will be performed by certified programs (i.e. SPSS, R). For risk stratification, conventional statistical methods, including Kaplan-Meier survival analysis, univariable and multivariable logistic regression, Cox regression model, and mixed models will be used. In addition, machine learning and artificial intelligence will be applied for the setting-up of cost-effective prediction models. The best indexes for descriptive statistics, as well as optimal tests for comparing quantitative and qualitative variables, will be chosen depending on the distribution of data, as appropriate. Confidence intervals will be set at 95%. Statistical significance threshold will be set at p <0.05 (two-sided).
Sampling Method: Probability Sample
Enrollment: 262 (Estimated)
Dates: Start 2025-02-25 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
To provide baseline characterization of VA in the study cohort. | Baseline
  Prevalence of baseline VA
To provide baseline characterization of VA in the study cohort. | baseline
  Type of VA
To provide baseline characterization of VA in the study cohort. | baseline
  Morphology of VA
To provide follow-up characterization of VA in study cohort. | 12 months
  Occurrence of VA by 12 months
To provide follow-up characterization of VA in study cohort. | 12 months
  Burden of VA (number of VA events per month)
To screen for CGVs in study groups | 6 months
  Prevalence of CGVs in myocarditis with VA (VA+) vs. without VA (VA-)
To screen for CGVs in study groups vs healthy controls | 6 months
  Prevalence of CGVs in myocarditis with VA (VA+) and without VA (VA-) vs. healthy controls
To investigate the pathophysiological basis of arrhythmic myocarditis in study group (exploratory endpoint) | during the procedure
  Comparison of gene expression profile on EMB in inflammatory group vs no inflammatory group

SECONDARY OUTCOMES:
To provide baseline characterization of VA according to sex | Baseline
  Prevalence of baseline VA in male vs female.
To provide baseline characterization of VA according to sex | baseline
  Type of VA in male vs female.
To provide baseline characterization of VA according to sex | baseline
  Morphology of VA in male vs female
To provide follow-up characterization of VA according to sex | 12 months
  Occurrence of VA by 12 months in male vs female.
To provide follow-up characterization of VA according to sex | 12 months
  Burden of VA (number of VA events per month) in male vs female.
To screen for CGVs in study groups | 6 months
  Prevalence of CGVs in myocarditis with VA (VA+) vs without VA (VA-)
To screen for CGVs in study groups vs healthy controls | 6 months
  Prevalence of CGVs in myocarditis with VA (VA+) and without VA (VA-) vs healthy controls
To investigate the pathophysiological basis of arrhythmic myocarditis according to sex (exploratory endpoint) | during the procedure
  Comparison of gene expression profile on EMB in inflammatory group vs no inflammatory group, in male vs female

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Della Bella, MD, Study Chair — Scientific Institute San Raffaele, Milan, Italy
Locations (1):
- Scientific Institute San Raffaele, Milan, Italy/Milan, Italy

REFERENCES:
- [Background] Tedesco M, Giannese F, Lazarevic D, Giansanti V, Rosano D, Monzani S, Catalano I, Grassi E, Zanella ER, Botrugno OA, Morelli L, Panina Bordignon P, Caravagna G, Bertotti A, Martino G, Aldrighetti L, Pasqualato S, Trusolino L, Cittaro D, Tonon G. Chromatin Velocity reveals epigenetic dynamics by single-cell profiling of heterochromatin and euchromatin. Nat Biotechnol. 2022 Feb;40(2):235-244. doi: 10.1038/s41587-021-01031-1. Epub 2021 Oct 11. PMID 34635836
- [Background] Tiron C, Campuzano O, Fernandez-Falgueras A, Alcalde M, Loma-Osorio P, Zamora E, Caballero A, Sarquella-Brugada G, Cesar S, Garcia-Cuenllas L, Garcia-Alvarez A, Jorda P, Arbelo E, Tomas-Querol C, Pineda V, Martinez D, Brugada R. Prevalence of Pathogenic Variants in Cardiomyopathy-Associated Genes in Myocarditis. Circ Genom Precis Med. 2022 Jun;15(3):e003408. doi: 10.1161/CIRCGEN.121.003408. Epub 2022 May 6. No abstract available. PMID 35522179
- [Background] Peretto G, Casella M, Merlo M, Benedetti S, Rizzo S, Cappelletto C, Di Resta C, Compagnucci P, De Gaspari M, Dello Russo A, Casari G, Basso C, Sala S, Sinagra G, Della Bella P, Cooper LT Jr. Inflammation on Endomyocardial Biopsy Predicts Risk of MACE in Undefined Left Ventricular Arrhythmogenic Cardiomyopathy. JACC Clin Electrophysiol. 2023 Jul;9(7 Pt 1):951-961. doi: 10.1016/j.jacep.2022.10.032. Epub 2023 Jan 18. PMID 36752457
- [Background] Richards S, Aziz N, Bale S, Bick D, Das S, Gastier-Foster J, Grody WW, Hegde M, Lyon E, Spector E, Voelkerding K, Rehm HL; ACMG Laboratory Quality Assurance Committee. Standards and guidelines for the interpretation of sequence variants: a joint consensus recommendation of the American College of Medical Genetics and Genomics and the Association for Molecular Pathology. Genet Med. 2015 May;17(5):405-24. doi: 10.1038/gim.2015.30. Epub 2015 Mar 5. PMID 25741868
- [Background] Peretto G, De Luca G, Villatore A, Di Resta C, Sala S, Palmisano A, Vignale D, Campochiaro C, Lazzeroni D, De Gaspari M, Rizzo S, Busnardo E, Ferro P, Gianolli L, Basso C, Dagna L, Esposito A, Benedetti S, Della Bella P. Multimodal Detection and Targeting of Biopsy-Proven Myocardial Inflammation in Genetic Cardiomyopathies: A Pilot Report. JACC Basic Transl Sci. 2023 Jul 5;8(7):755-765. doi: 10.1016/j.jacbts.2023.02.018. eCollection 2023 Jul. PMID 37547072
- [Background] Peretto G, Sala S, Basso C, Rizzo S, Radinovic A, Frontera A, Limite LR, Paglino G, Bisceglia C, De Luca G, Campochiaro C, Sartorelli S, Palmisano A, Esposito A, Busnardo E, Villatore A, Baratto F, Cireddu M, Marzi A, D'Angelo G, Gulletta S, Vergara P, De Cobelli F, Dagna L, Mazzone P, Della Bella P. Inflammation as a Predictor of Recurrent Ventricular Tachycardia After Ablation in Patients With Myocarditis. J Am Coll Cardiol. 2020 Oct 6;76(14):1644-1656. doi: 10.1016/j.jacc.2020.08.012. PMID 33004129
- [Background] Peretto G, Sala S, De Luca G, Marcolongo R, Campochiaro C, Sartorelli S, Tresoldi M, Foppoli L, Palmisano A, Esposito A, De Cobelli F, Rizzo S, Thiene G, Basso C, Dagna L, Caforio ALP, Della Bella P. Immunosuppressive Therapy and Risk Stratification of Patients With Myocarditis Presenting With Ventricular Arrhythmias. JACC Clin Electrophysiol. 2020 Oct;6(10):1221-1234. doi: 10.1016/j.jacep.2020.05.013. Epub 2020 Jun 24. PMID 33092747
- [Background] Peretto G, Sala S, Rizzo S, Palmisano A, Esposito A, De Cobelli F, Campochiaro C, De Luca G, Foppoli L, Dagna L, Thiene G, Basso C, Della Bella P. Ventricular Arrhythmias in Myocarditis: Characterization and Relationships With Myocardial Inflammation. J Am Coll Cardiol. 2020 Mar 10;75(9):1046-1057. doi: 10.1016/j.jacc.2020.01.036. PMID 32138965
- [Background] Mantri M, Hinchman MM, McKellar DW, Wang MFZ, Cross ST, Parker JSL, De Vlaminck I. Spatiotemporal transcriptomics reveals pathogenesis of viral myocarditis. Nat Cardiovasc Res. 2022 Oct;1(10):946-960. doi: 10.1038/s44161-022-00138-1. Epub 2022 Oct 10. PMID 36970396
- [Background] Rizzo S, Lodder EM, Verkerk AO, Wolswinkel R, Beekman L, Pilichou K, Basso C, Remme CA, Thiene G, Bezzina CR. Intercalated disc abnormalities, reduced Na(+) current density, and conduction slowing in desmoglein-2 mutant mice prior to cardiomyopathic changes. Cardiovasc Res. 2012 Sep 1;95(4):409-18. doi: 10.1093/cvr/cvs219. Epub 2012 Jul 3. PMID 22764152
- [Background] Vermij SH, Abriel H, van Veen TA. Refining the molecular organization of the cardiac intercalated disc. Cardiovasc Res. 2017 Mar 1;113(3):259-275. doi: 10.1093/cvr/cvw259. PMID 28069669
- [Background] Ammirati E, Raimondi F, Piriou N, Sardo Infirri L, Mohiddin SA, Mazzanti A, Shenoy C, Cavallari UA, Imazio M, Aquaro GD, Olivotto I, Pedrotti P, Sekhri N, Van de Heyning CM, Broeckx G, Peretto G, Guttmann O, Dellegrottaglie S, Scatteia A, Gentile P, Merlo M, Goldberg RI, Reyentovich A, Sciamanna C, Klaassen S, Poller W, Trankle CR, Abbate A, Keren A, Horowitz-Cederboim S, Cadrin-Tourigny J, Tadros R, Annoni GA, Bonoldi E, Toquet C, Marteau L, Probst V, Trochu JN, Kissopoulou A, Grosu A, Kukavica D, Trancuccio A, Gil C, Tini G, Pedrazzini M, Torchio M, Sinagra G, Gimeno JR, Bernasconi D, Valsecchi MG, Klingel K, Adler ED, Camici PG, Cooper LT Jr. Acute Myocarditis Associated With Desmosomal Gene Variants. JACC Heart Fail. 2022 Oct;10(10):714-727. doi: 10.1016/j.jchf.2022.06.013. Epub 2022 Sep 7. PMID 36175056
- [Background] Peretto G, Sala S, Rizzo S, De Luca G, Campochiaro C, Sartorelli S, Benedetti G, Palmisano A, Esposito A, Tresoldi M, Thiene G, Basso C, Della Bella P. Arrhythmias in myocarditis: State of the art. Heart Rhythm. 2019 May;16(5):793-801. doi: 10.1016/j.hrthm.2018.11.024. Epub 2018 Nov 24. PMID 30476544
- [Background] Peretto G, Sommariva E, Di Resta C, Rabino M, Villatore A, Lazzeroni D, Sala S, Pompilio G, Cooper LT. Myocardial Inflammation as a Manifestation of Genetic Cardiomyopathies: From Bedside to the Bench. Biomolecules. 2023 Apr 4;13(4):646. doi: 10.3390/biom13040646. PMID 37189393
- [Background] Caforio AL, Pankuweit S, Arbustini E, Basso C, Gimeno-Blanes J, Felix SB, Fu M, Helio T, Heymans S, Jahns R, Klingel K, Linhart A, Maisch B, McKenna W, Mogensen J, Pinto YM, Ristic A, Schultheiss HP, Seggewiss H, Tavazzi L, Thiene G, Yilmaz A, Charron P, Elliott PM; European Society of Cardiology Working Group on Myocardial and Pericardial Diseases. Current state of knowledge on aetiology, diagnosis, management, and therapy of myocarditis: a position statement of the European Society of Cardiology Working Group on Myocardial and Pericardial Diseases. Eur Heart J. 2013 Sep;34(33):2636-48, 2648a-2648d. doi: 10.1093/eurheartj/eht210. Epub 2013 Jul 3. PMID 23824828